CLINICAL TRIAL: NCT03625804
Title: The Motor Effects of Combined Peripheral Nerve Electrical Stimulation and Action Observation on the Affected Hand in People With Stroke
Brief Title: The Cortical Motor Effects of PNS and AO on Motor Training in Chronic Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LIU Hao, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20140617001-01
Record Dates: First submitted 2018-06-28; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Stroke
Keywords: Electrical Stimulation; Cortical Excitability; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: Single-blind randomized cross-over study
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PNS+AO+Training (Experimental): adopted "PNS+AO+Training" as the intervention
  Interventions: Genetic: PNS+AO+Training
- PNS+AOsham+Training (Experimental): adopted "PNS+AOsham+Training" as the intervention
  Interventions: Genetic: PNS+AOsham+Training
- PNSsham+AOsham+Training (Placebo Comparator): adopted "PNSsham+AOsham+Training" as the intervention
  Interventions: Genetic: PNSsham+AOsham+Training

INTERVENTIONS:
Genetic: PNS+AO+Training — Electrical stimulation was applied to the radial and ulnar nerve (PNS) of the paretic arm for 60 minutes. During the last 30 minutes of PNS, action observation (AO) was introduced in which subjects were required to watch a series of video clips. After one hour's PNS+AO, the subjects then proceeded to a 30-minute period of motor training of paretic hand.
  Arms: PNS+AO+Training
Genetic: PNS+AOsham+Training — PNS was given as described before. During the last 30 minutes of the PNS, subjects were shown different photos illustrating a letter, a number or a hand as AOsham. The protocol of motor training was the same as described before.
  Arms: PNS+AOsham+Training
Genetic: PNSsham+AOsham+Training — The 1-hour PNSsham was conducted with the electrical stimulation unit turned on but without current output. The protocols for AOsham and motor training were the same as those described before.
  Arms: PNSsham+AOsham+Training

SUMMARY:
This study aimed to investigate if peripheral nerve stimulation (PNS) paired with action observation (AO) would augment motor training in promoting corticomotor excitability for the paretic hand in people with stroke. Twenty subjects in chronic stage of stroke were exposed to 3 different interventions involving one-hour PNS or sham PNS paired with 30 minutes of AO or sham AO, all followed by 30 minutes of finger abduction training in 3 separate sessions.

DETAILED DESCRIPTION:
The investigator's previous study (Liu & Au-Yeung, 2017; PMID: 28383292) has demonstrated that 1-hour peripheral nerve stimulation (PNS) applied to the radial and ulnar nerves of the paretic UL of people with chronic stroke can increase transcranial magnetic stimulation (TMS)-evoked excitability of corticomotor pathways in both hemispheres projected to the contralateral first dorsal interosseous (FDI) hand muscle, and also improve dexterity in the paretic hand. This bi-hemispheric effect of PNS suggests that certain additional therapies such as action observation (AO) and motor training should be incorporated to strengthen the plastic corticomotor adaptation specifically for paretic UL control. The hypothesis of this study is that PNS paired with AO would augment task training of the paretic hand by increasing the corticomotor excitability in the lesioned hemisphere for the trained hand muscle in people with stroke, with associated dexterity function improvement. Twenty subjects were recruited by convenience in the community. They then attended an assessment session to evaluate the baseline sensorimotor status of their paretic upper limb. After the clinical tests，the subjects were introduced the assessment procedure for measuring corticomotor excitability with transcranial magnetic stimulation (TMS). After 1-week intermission, the subjects returned for 3 intervention sessions with different protocols including (1)PNS+AO+Training; (2)PNS+AOsham+Training; and (3)PNSsham+AOsham+Training. These 3 intervention sessions were arranged in random sequence for subjects. For "PNS+AO+Training" session, electrical stimulation was applied to the radial and ulnar nerve (PNS) of the paretic arm for 60 minutes. During the last 30 minutes of PNS, action observation (AO) was introduced in which subjects were required to watch a series of video clips. After one hour's PNS+AO, the subjects then proceeded to a 30-minute period of motor training of paretic hand. During "PNS+AOsham+Training" session, PNS was given as described before. During the last 30 minutes of the PNS, subjects were shown different photos illustrating a letter, a number or a hand as AOsham. The protocol of motor training was the same as described before. In the session of "PNSsham+AOsham+Training", The 1-hour PNSsham was conducted with the electrical stimulation unit turned on but without current output. The protocols for AOsham and motor training were the same as those described before.

ELIGIBILITY:
Inclusion Criteria:

* age between 40 and 80 years;
* has history of first hemispheric stroke of 6or more months;
* presence of electromyographic signals in first dorsal interosseous (FDI) during active abduction of the index finger contralateral to the lesioned hemisphere;
* medically stable;
* able to comprehend instructions.

Exclusion Criteria:

* past history of musculoskeletal or neurological impairment in the paretic upper limb;
* recurrent stroke;
* cognitive impairment (Mini-mental state examination (MMSE) < 24);
* visual impairment not correctable by optical lens;
* presence of metal in the head region or a cardiac pacemaker as contraindications for TMS (Rossi et al., 2009).

Ages: 43 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-06-23 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Corticomotor excitability evoked by Transcranial magnetic stimulation (TMS) | 90 minutes
  Corticomotor excitability in terms of the slope of the MEP recruitment curve and peak MEP amplitude captured for the contralateral FDI hand muscle in both hemispheres were assessed.

SECONDARY OUTCOMES:
Hand dexterity of paretic hand evaluated with Purdue Pegboard | 24 hours
  The score was the total number of pins inserted into the holes with paretic hand in 30 seconds.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2014-10-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03625804/ICF_000.pdf